CLINICAL TRIAL: NCT00299403
Title: The Antidepressant Effect of Repetitive Transcranial Magnetic Stimulation (rTMS)Compared to Electroconvulsive Therapy (ECT).An Open Randomized Noninferiority Trial.
Brief Title: The Antidepressant Effect of Repetitive Transcranial Magnetic Stimulation (rTMS)Compared to ECT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Poul Erik Buchholtz Hansen, Aarhus University Hospital , Risskov. Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20010072
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Depressive Disorder
Keywords: Depressive disorder,; Antidepressant effect,; rTMS,; ECT,; cognition,; Saliva cortisol; noninferiority trial
MeSH Terms: conditions — Depressive Disorder | interventions — Transcranial Magnetic Stimulation; Electroconvulsive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Right frontal low frequency rTMS
  Interventions: Procedure: Right prefrontal lowfrequency ( 1 hz) rTMS.
- 2 (Active Comparator): electroconvulsive therapy (ECT). Right unilateral ECT 3 time a week in 3 weeks
  Interventions: Procedure: Electroconvulsive therapy (ECT)

INTERVENTIONS:
Procedure: Right prefrontal lowfrequency ( 1 hz) rTMS. — Right prefrontal low frequency (1 hz) rTMS. 15 sessions with one daily session during 3 weeks (weekends excluded). Each session covering 2 x 60 minutes of stimulation separated with an intertrain interval of 3 minutes
  Arms: 2
  Arms: 1
Procedure: Electroconvulsive therapy (ECT) — 9 ECT ( 3 each week) during 3 weeks
  Arms: 2

SUMMARY:
The aim of the present study is to compare the antidepressant effect of electroconvulsive therapy ( ECT) with that of low frequency repetitive transcranial magnetic stimulation of the right prefrontal cortex.

In the same study we investigate the value of saliva cortisol as a predictor of treatment outcome.

DETAILED DESCRIPTION:
Previous clinical controlled trials indicate that repetitive transcranial magnetic stimulation (rTMS) of the prefrontal cortex may relieve antidepressant symptoms. Most of these studies have used high frequency stimulation of the left frontal cortex. A few investigations have found that right frontal low frequency rTMS, which constitute a more gentle stimulus design has an antidepressant effective at the same level. Compared to ECT rTMS has obvious advantages. The new method implies focal stimulation of the brain, is not inducing epileptic seizures and does not require anesthesia. In addition rTMS does not seem to induce cognitive disturbances. Few studies have compared the antidepressant effect of rTMS with that of ECT. The main outcome indicates that high frequency rTMS of the left frontal cortex has an antidepressant effect which is comparable to that of ECT in the treatment of non-psychotic patients. It is difficult to draw definite conclusions from these studies, first of all because of small and highly selected study populations. In addition different stimulus designs make most of the mentioned studies incomparable.

The aim of the present study is to compare the antidepressant effect of low frequency rTMS of the right dorsolateral prefrontal cortex with ECT in a hospitalized population of major depressed patients (ICD-10/DSM-IV) in a randomized open noninferiority study.

About fifty percent of depressed patients have shown to be associated with an increased plasma cortisol concentration and HPA-axis activity expressed in non-suppression of plasma cortisol in association with the dexamethasone (DX-test) suppression test. Some studies have shown that the presence or absence of normalization of the HPA-axis activity and the DX-test during antidepressant treatment may be a predictor of recurrence. Other studies have shown that the physiological increase in the concentration of saliva cortisol during the first half an hour after awakening in the morning is accentuated in depressed patients and constitute a more simple expression of the HPA-.axis activity and predictor of outcome than the the dx-test.

Therefore we want to investigate the value of the increase in the morning cortisol concentration during the first half an hour after awakening as a predictor of antidepressant effect and outcome.

ELIGIBILITY:
Inclusion Criteria

* Admission to Psychiatric Hospital in Aarhus.
* The patient should be candidate for ECT.
* Moderate or severely depressed/Major depressed (ICD-10/DSM-IV)
* A total score on the Hamilton (17-item) rating scale for depression of 20 or above, or a subscale score of 10 ore above.
* Right handed,
* Age 18-80 years

Exclusion Criteria:

* Organic brain disease
* Epilepsy
* Metal devices in operated into the brain or chest.
* The patient is wearing cardiac pacemaker.
* Medical illness associated with disturbed CNS function
* Pregnancy
* Serious suicidality
* Severe agitation or delirium
* Alcoholic or drug dependency
* The patients exposed to coercive measures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The total 17-item score on the Hamilton Rating Scale for depression | during 3 weeks of treatment and 4 week s after last treatment

SECONDARY OUTCOMES:
UKU-side effect score | at baseline at day 10 during the treatment period, just after termination of treatment and after 4 weeks of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Poul Erik Buchholtz Hansen, senior phys., Principal Investigator — Aarhus University Hospital, Risskov, Denmark
Locations (1):
- University hospital of Aarhus, Risskov, Aarhus, Risskov, Denmark

REFERENCES:
- [Background] Klein E, Kreinin I, Chistyakov A, Koren D, Mecz L, Marmur S, Ben-Shachar D, Feinsod M. Therapeutic efficacy of right prefrontal slow repetitive transcranial magnetic stimulation in major depression: a double-blind controlled study. Arch Gen Psychiatry. 1999 Apr;56(4):315-20. doi: 10.1001/archpsyc.56.4.315. PMID 10197825
- [Derived] Hansen PE, Ravnkilde B, Videbech P, Clemmensen K, Sturlason R, Reiner M, Parner E, Rosenberg R, Vestergaard P. Low-frequency repetitive transcranial magnetic stimulation inferior to electroconvulsive therapy in treating depression. J ECT. 2011 Mar;27(1):26-32. doi: 10.1097/YCT.0b013e3181d77645. PMID 20351570